CLINICAL TRIAL: NCT01961323
Title: Effects of Nebivolol on Left Ventricular and Left Atrial Morphodynamics in Adults With Hypertension and Isolated Diastolic Dysfunction
Brief Title: Effect of Nebivolol on the Blood Flow in Hearts of Adults With High Blood Pressure and Abnormal Filling of Heart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Partho Sengupta, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0493
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Hypertension; Left Ventricular Diastolic Dysfunction
Keywords: Hypertension; high blood pressure; stress echocardiogram; nebivolol; left ventricular diastolic dysfunction
MeSH Terms: conditions — Hypertension; Ventricular Dysfunction, Left | interventions — Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nebivolol (Experimental): Nebivolol 5 mg (titrated to a maximal dose of 10mg for optimal blood pressure) for 6 months
  Interventions: Drug: Nebivolol

INTERVENTIONS:
Drug: Nebivolol — Doses will be titrated based on weekly visits during the first 2 weeks to achieve a target SBP<140 and DBP <90 mm Hg. If BP remains uncontrolled after 2 weeks of treatment, indapamide will be added at a dosage of 2.5 mg/day. If the therapeutic goal is still not achieved by 4 weeks, patients will be withdrawn from the study.Upward titration will be halted, and the previous dosage level resumed, if at any point systolic blood pressure falls to ≤ 100 mmHg, even if the individual remains asymptomatic.

SUMMARY:
To investigate whether treatment with Nebivolol in subjects with high blood pressure and abnormal filling of left ventricle (LVDD) improves exercise time by improving Left Ventricular deformation and filling.

DETAILED DESCRIPTION:
Background:

The left ventricle (LV) ejects blood with a wringing motion, where the LV apex rotates counterclockwise and the base rotates in clockwise directions respectively. Rapid untwisting and recoil of LV during isovolumic relaxation and early diastole releases energy stored in ejection for LV suction and rapid early diastolic restoration. The LV geometry and its rotational mechanics also give rise to intracavitary blood flow rotation resulting into LV intracavitary vortex ring formation. LV torsion and vortex ring formation confer morphodynamic advantages that gain importance as blood flow velocities, heart rate and rates of change of momentum increase with exertion for improving LV efficiency. We have recently characterized the significance of LV twist mechanics and vortex ring formation in human hearts using novel high resolution speckle and contrast particle tracking echocardiography. Although data on a favorable effect of nebivolol on exercise capacity and LV diastolic filling exists, the changes in left ventricular (LV) rotational mechanics and blood flow vortex ring formation that may explain the potential hemodynamic benefits seen with nebivolol have not been previously characterized.

Aims:

In patients with hypertension and left ventricular diastolic dysfunction (LVDD) treatment with nebivolol for 6 months improves exercise time by enhancing:

1. LV deformation, torsion and untwisting mechanics
2. LA-to-LV blood flow transport and characteristics of intra-cavitary vortex formation
3. LA reservoir and booster pump function and LA-LV interaction during the conduit phase

Hypotheses:

Treatment with nebivolol in subjects with hypertension and LVDD improves exercise time by improving LV deformation and diastolic filling. As diastole shortens with the tachycardia associated with exercise, the contribution of untwist becomes relatively more important to LV suction and filling. Nebivolol improves LV diastolic filling primarily by enhancing LV untwisting and the rheological efficiency of blood flow transport through vortex formation in early diastole.

Significance:

Patients with LVDD are asymptomatic at rest and often but become markedly symptomatic with exertion. This pilot study will provide data for the first time for correlating the improvement in exercise capacity seen with the use of nebivolol with the changes in LV relaxation, torsional mechanics, LV vortex formation and LA-LV transport functions. The preliminary data will be essential for understanding the underlying pathophysiological mechanisms through which nebivolol improves exercise hemodynamics besides providing data for development of subsequent larger randomized multicentric trials.

ELIGIBILITY:
Inclusion Criteria:

* History of mild (140-160 / 90-100) to moderate (160-200 / 100-120) hypertension
* LV diastolic dysfunction (>/= Grade1)
* LV ejection fraction >50%
* Indexed left atrial volume >/= 28 mL/m^2
* In sinus rhythm at the time of enrollment
* Willingness to return for the 6-month follow up investigations

Exclusion Criteria:

* Presence or history of any of the following at baseline:

  1. History of mitral valve disease of greater than mild severity or prosthetic mitral valve, congenital heart disease or permanent pacemaker
  2. Calculated creatinine clearance <50 mL/min
  3. Terminal Illness with expected Survival of <1 year
  4. Previous Heart Transplant
  5. Individuals who are institutionalized
  6. Systolic BP>180 mm Hg or diastolic BP > 120 mm Hg
* Medical treatment for elevated BP with:

  1. Calcium channel blocker (e.g. verapamil, nifedipine);
  2. Alpha blocker (e.g. prazosin);
  3. Alpha agonist (e.g. α-methyldopa, hydralazine, clonidine)
* Patient unwilling or unable to provide informed consent for study participation
* Pregnancy (current, or anticipated within the study period)
* Secondary Hypertension
* Previous echo contrast allergy
* Poor echocardiography window
* Previous stroke, known carotid stenosis
* Contraindication for beta-blocker therapy (sinus bradycardia <50 beats/min);
* 2nd or 3rd degree AV conduction block
* Overt congestive cardiac failure (NYHA Class III-IV)
* Known bronchospastic disease
* Known hepatic dysfunction (SGOT/PT > twice above normal levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partho Sengupta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Icahn School of Medicine at Mount Sinai outpatient cardiology clinic from Dec 11, 2014 to Dec 2, 2016.
Groups:
- Nebivolol: Nebivolol 5 mg (titrated to a maximal dose of 10mg for optimal blood pressure) for 6 months
  Nebivolol: Doses titrated based on weekly visits during the first 2 weeks to achieve a target SBP<140 and DBP <90 mm Hg. If BP remains uncontrolled after 2 weeks of treatment, indapamide will be added at a dosage of 2.5 mg/day. If the therapeutic goal is still not achieved by 4 weeks, patients will be withdrawn from the study.Upward titration will be halted, and the previous dosage level resumed, if at any point systolic blood pressure falls to ≤ 100 mmHg, even if the individual remains asymptomatic.
Period: Overall Study
Arm/Group | Nebivolol
Started | 70
Completed | 21
Not Completed | 49
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 8
Not completed — screen failure | 34

BASELINE CHARACTERISTICS:
Arm/Group | Nebivolol
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31 (6.6)
B-type Natriuretic Peptide (BNP) Blood Test [Mean (Standard Deviation); unit: pg/mL] — B-type natriuretic peptide (BNP) is a hormone produced by the heart. It is released in response to changes in pressure inside the heart. In general, the level of BNP goes up when heart failure develops or gets worse, and it goes down when the condition is stable.
  pg/mL | 19.8 (13)
Resting Heart Rate [Mean (Standard Deviation); unit: beat/minute] | 74.5 (14)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHG] | 142 (16.6)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHG] | 92.9 (10)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Exercise Tolerance
Description: measured by stress echocardiogram, number of participants who had improvement in METS and improvement in exercise time as compared to their baseline.
Time Frame: at 6 months
Population: Study results only for those who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 21
Participants
  Improvement in METs and exercise time | 9
  Improvement in exercise time only | 8

2. Secondary Outcome: E Velocity Indexed to e' (E/e' Ratio) of the Left Ventricle
Description: measured as a part of stress echocardiogram, E/e' ratio: The normal E/e' ratio from the medial annulus is <8 and suggests a normal left atrial pressure. While values between 8 and 12 are indeterminate, a value >12 is indicative of an elevated left atrial pressure or PCWP (>18mmHg). The ranges for E/e' from the lateral mitral annulus are <5, 5 -10 and >10 respectively.
Time Frame: at 6 months
Population: Results for the participants who had improved exercise capacity only (from Outcome Measure 1)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nebivolol
Number analyzed (Participants) | 17
ratio
  Resting | 7.5 (5.2)
  Peak Exercise | 8.8 (1.6)

3. Secondary Outcome: Untwist Rate of the Left Ventricle
Description: measured as a part of stress echocardiogram, number of participants with significant improvement in the LV untwist after Nebivolol treatment in patients who completed the study
Time Frame: at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nebivolol
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Arm/Group | Nebivolol
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No